CLINICAL TRIAL: NCT03428568
Title: Open Label, Randomized, Single Site Clinical Trial To Compare The Safety Of Herbal Melanin Extracted From Nigella Sativa Seeds Vs Standard Of Care Treatment In Treating Gastritis Patients
Brief Title: Safety Trial of Herbal Melanin in Gastritis Patients
Acronym: RASATHEME
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King Abdullah International Medical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC15/152/R
Record Dates: First submitted 2018-01-14; First posted 2018-02-09 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2017-12

CONDITIONS: Acid Dyspepsia; Gastritis
Keywords: Herbal Melanin; H.Pylori
MeSH Terms: conditions — Gastritis | interventions — Esomeprazole; Amoxicillin; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Herbal Melanin (Experimental): Herbal melanin 1800 milligram(mg) orally thrice a day with meals (300mgx2 capsules)
  Interventions: Other: Herbal Melanin
- Nexium (Active Comparator): omeprazole 40 mg once per day for one month.
  Interventions: Drug: Nexium
- H-Pylori infected : Herbal Melanin (Experimental): Herbal melanin 1800 mg orally thrice a day(TID) with meals (300 mg x2 capsules)
  Interventions: Other: Herbal Melanin
- nexium+ amoxil+clarithromycin (Active Comparator): omeprazole40 mg P.O. Twice per Day(BID) for one month + Amoxil 1000mg P.O. BID for 2 weeks+ Clarithromycin500 mg PO BID for two weeks.
  Omeprazole+Amoxil+clarithromycin is the standard triple therapy given
  Interventions: Drug: Nexium; Drug: Amoxil; Drug: Clarithromycin
- nexium +Herbal melanin (Experimental): omeprazole 40 mg P.O. BID for one month +1800 mg Herbal melanin PO TID (300mg x2 capsules) Omeprazole + Herbal melanin will be tested
  Interventions: Other: Herbal Melanin; Drug: Nexium
- Herbal melanin+amoxil+ clarithromycin (Experimental): Amoxil 1000mg P.O. BID for 2 weeks+ Clarithromycin500 mg PO BID for two weeks +1800 mg Herbal melanin PO TID(300 mg X 2 capsules) Herbal melanin+Amoxil+Clarithromycin will be tested
  Interventions: Other: Herbal Melanin; Drug: Amoxil; Drug: Clarithromycin

INTERVENTIONS:
Other: Herbal Melanin — Herbal melanin extracted from Nigella sativa seeds
  Other Names: Melanole
  Arms: H-Pylori infected : Herbal Melanin; Herbal Melanin; Herbal melanin+amoxil+ clarithromycin; nexium +Herbal melanin
Drug: Nexium — omeprazole
  Other Names: Aciloc
  Arms: Nexium; nexium +Herbal melanin; nexium+ amoxil+clarithromycin
Drug: Amoxil — Antibiotic
  Arms: Herbal melanin+amoxil+ clarithromycin; nexium+ amoxil+clarithromycin
Drug: Clarithromycin — Antibiotic
  Other Names: Klacid
  Arms: Herbal melanin+amoxil+ clarithromycin; nexium+ amoxil+clarithromycin

SUMMARY:
The aim of the study is to use Melanole, a herbal extract from Nigella sativa, for treatment of gastritis. The effect of Melanole will be compared between participants (including H. pylori and non-H.pylori infected patients), with the triple therapy and Standard of care treatment of gastritis, respectively.

All participants will be examined before and after the administration of Melanole. The results showing a relief of gastritis symptoms for non-H. pylori patients and partial or complete eradication of H. pylori for H.pylori infected patients will be evaluated.

DETAILED DESCRIPTION:
Background:

The melanin to be used in this study is a herbal melanin (HM) that has been extracted from the plant Nigella sativa. Nigella sativa was obtained from local market in Riyadh, Saudi Arabia. HM has been obtained from seed total powdered extract using standard extraction procedure and has been reported as a patent for the first time.The percentage of pure melanin in total Nigella sativa L. is 9% as identified using Electron Spin Resonance (ESR) and Fourier Transform- Infra Red (FI-IR) and calculated using wet chemical methods. Three different patches of Nigella sativa L that were obtained from different Nigella sativa L species were tested (Saudi, Ethiopian and Indian) and the same percentage of HM was obtained. The safety of HM has been tested and confirmed by different labs including lab for Quality and Safety and Industrial Research Institute(IRI) (see supplements 1 and 2). Similarly, the safety of the HM capsules have been tested at the Toxicology and Bioanalysis in King Faisal Specialist Hospital(KFSH) (see supplement 3). Moreover, the capsules have been approved and certified for free sale by the Ministry of Health at Lebanon.

Study Area:

The study will be performed in the gastroenterology clinic at National Guard Health Affairs(NGHA). Volunteers who participate in the study will be recruited from NGHA clinics. Participates are patients diagnosed with gastritis, both H. Pylori and non-H.Pylori infected, together with healthy volunteers.

The histological studies will be performed at the pathology department at NGHA.

Taking biopsies during endoscopy:

The best way to get tissue samples from the stomach is through a procedure called an esophagogastroduodenoscopy. It is more commonly known as an endoscopy or EGD. This is generally done as an outpatient procedure. The biopsies will be taken through the esophagogastroduodenoscopy (EGD) by a ultra-thin forceps, then will be saved in special container and send to the Laboratory for staining and microscopic examination. Under the microscope the pathologist will look for the abnormal mucosa , inflammation, ulceration , and helicobacter pylori gram negative micro-organism .During the procedure there is low chance of some complications which happened in 1: 10 000 , these include ; injury to the mucosa with bleeding and perforation , discomfort , sedation related complication like headache and nausea . These rare but the patient will be informed about it.

Study Subjects:

Patients with gastritis or showing gastritis symptoms will be enrolled in this study. Gastritis participate patients will be selected after detection of gastric lesions by undergoing routine diagnostic tests (such as endoscopy of upper digestive system).

Sample Size Calculation and Estimation:

The sample size has been estimated as 132 ( 22 subjects per group). The calculation and estimation have been done as follows:

Sample Size Calculation

The calculation of sample size was performed using Query Advisor V.7

Sample Size Estimated

The minimum number of Subjects needed in each group is 18, a two sided 95.0% confidence interval for the difference between a Group 1 proportion of 0.6 and Group 2 proportion of 0.2 based on the large sample normal approximation will extend 0.3 from the observed differences in proportions. The total required sample would be (6 groups x 18=108).The assumed withdrawal/dropout rate is 20% in each group (22 subjects per group), the final sample size would ne 132 subjects. The calculation of sample size was performed using Query Advisor V.7)

Data Collection method:

All data will be collected electronically and reported in Case Report Forms.

Data Cleaning:

Raw data will be processed in accordance with the best practices for raw data management to identify any inaccuracies or incompleteness in advance to the statistical analysis. In order to accomplish this task, all interval variables will be checked and summarized in terms of maximum and minimum values. Minimum and maximum values will be checked and compared against the nominal maximum and minimum value of each variable and variables with implausible values will be flagged. A similar process will be applied to categorical variables to identify any potential anomalies (miscode) by running a general frequency analysis.

Cohort Characterization:

All variables will be summarized and reported using descriptive statistics. Interval variables will be summarized and reported in terms of mean and standard deviation. Categorical variables will be summarized and reported in terms of frequency distribution. All variables will be compared across study groups using chi square and t test accordingly.

Primary Outcome(s) Analysis:

Chi square test will be used to compare the distribution of gastritis across the study groups. Results will be reported in terms of count, percent, and p-value. Significance will be declared at alfa less than 0.05. Binary logistic regression will be used to identify significant predictors of the primary outcomes. The statistical model will include key variables that showed significance with the primary outcome at the bivariate level. Results will be reported in terms of odds ratio, std. error, 95% confidence interval, and p-value. Significance will be declared at alfa less than 0.05.

Intent to treat analysis will be the approach in analyzing the data.

Statistical Analytical System(SAS) 9.2 will be used for all statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* Males or Females between 18- 60 years
* Willing to sign Informed Consent Form (ICF)
* Women of Child bearing age will be asked to conduct a pregnancy test before enrolling in the study and offered contraceptives for the duration of the study participation
* Clinical Pictures of Gastritis.
* Histologically confirmed H- Pylori Gastritis or Non H- Pylori by one week from enrollment.

Exclusion Criteria:

* Patients with disturbed gastrointestinal physiology (gastric surgery, vagotomy, Zollinger-Ellison syndrome)
* Patients who have been treated with proton pump inhibitors during 3 weeks prior to inclusion
* Patients who have been treated with antibiotics or bismuth containing drugs 1 month prior enrolling in the study
* Patient with pyloric stenosis
* Patient with Hematologic disorder
* Patient with congestive heart disease
* Women who are pregnant or lactating
* Current or past history of malignancy
* Drug abuser and chronic alcoholism
* Patients currently participating in any other clinical trial of any kind

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 132 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants cured from acidity symptoms and H.Pylori -induced gastritis | 6 months
  Investigators hypothesize that HM is an effective candidate that can decrease stomach acidity and eradicate H.Pylori by working as Proton Pump Inhibitor(PPI) and/or antibacterial agent, respectively. Investigators suggest the role of HM in activation of Toll like Receptor 4 (TLR4)/Cycloxygenase2(COX2)/ProstaglandinE2( PGE2) as one underlying mechanism.

SECONDARY OUTCOMES:
Number of Participants cured with herbal melanin as compared to number of participants cured with standard of care for gastritis and H.Pylori-induced gastritis | 6 months
  Gastritis as indicated by improving the clinical presentation of gastritis and confirmed by end of treatment endoscopy and stool antigen test
Number of Participants between study groups having high expression of TLR4 and COX2 as assessed by Western blots procedure. | 6 months
  By using stomach biopsies for measuring the expression of TLR4 and COX 2 expression.

CONTACTS AND LOCATIONS:
Overall Officials: Adila SA Elobeid, PhD, Principal Investigator — Ministry of National Guard

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] El-Obeid A, Al-Harbi S, Al-Jomah N, Hassib A. Herbal melanin modulates tumor necrosis factor alpha (TNF-alpha), interleukin 6 (IL-6) and vascular endothelial growth factor (VEGF) production. Phytomedicine. 2006 May;13(5):324-33. doi: 10.1016/j.phymed.2005.03.007. Epub 2005 Sep 19. PMID 16635740
- [Background] Biotechnological Method for Production of Melanin Pigments. Patent, award by Swedish PRV Patent office-Stockholm 2011 and United Nations PCT-WIPO 2011. Registered in US &Canada
- [Background] Extraction of melanin from Nigella sativa L. Patent No. 451, Khartoum, Sudan. 1998.
- [Background] Tortora, G.J. and Grabowski, S.R. (2003). Principles of Anatomy and Physiology. 10th ed. John Wiley& Sons, Inc, NJ, p.889.).
- [Background] Parkin DM. International variation. Oncogene. 2004 Aug 23;23(38):6329-40. doi: 10.1038/sj.onc.1207726. PMID 15322508
- [Background] Peleteiro B, Bastos A, Ferro A, Lunet N. Erratum to: Prevalence of Helicobacter pylori Infection Worldwide: A Systematic Review of Studies with National Coverage. Dig Dis Sci. 2015 Sep;60(9):2849. doi: 10.1007/s10620-015-3779-5. No abstract available. PMID 26160435
- [Background] Ayala G, Escobedo-Hinojosa WI, de la Cruz-Herrera CF, Romero I. Exploring alternative treatments for Helicobacter pylori infection. World J Gastroenterol. 2014 Feb 14;20(6):1450-69. doi: 10.3748/wjg.v20.i6.1450. PMID 24587621
- [Background] Hawkins C, Hanks GW. The gastroduodenal toxicity of nonsteroidal anti-inflammatory drugs: a review of the literature. J Pain Symptom Manage. 2000 Aug;20(2):140-51. doi: 10.1016/s0885-3924(00)00175-5. PMID 10989252
- [Background] El-Tahir, K. E. H.; Hassib, A. M.; El-Hag, H.; Ponten, F.; Westermark, B. El- Obeid Adila (2009). Anti-ulcerogenic effects of Nigella sativa Melanin. Sudan Patent No. 1683.
- [Background] Mimura T, Maeda K, Tsujibo H, Satake M, Fujita T. Studies on biological activities of melanin from marine animals. II. Purification of melanin from Octopus vulgaris Cuvier and its inhibitory activity on gastric juice secretion in rats. Chem Pharm Bull (Tokyo). 1982 Apr;30(4):1508-12. doi: 10.1248/cpb.30.1508. No abstract available. PMID 7105266
- [Background] Mimura T, Maeda K, Terada T, Oda Y, Morishita K, Aonuma S. Studies on biological activities of melanin from marine animals. III. Inhibitory effect of SM II (low molecular weight melanoprotein from squid) on phenylbutazone-induced ulceration in gastric mucosa in rats, and its mechanism of action. Chem Pharm Bull (Tokyo). 1985 May;33(5):2052-60. doi: 10.1248/cpb.33.2052. No abstract available. PMID 4053227
- [Background] El-Dakhakhny M, Barakat M, El-Halim MA, Aly SM. Effects of Nigella sativa oil on gastric secretion and ethanol induced ulcer in rats. J Ethnopharmacol. 2000 Sep;72(1-2):299-304. doi: 10.1016/s0378-8741(00)00235-x. PMID 10967486
- [Background] Kanter M, Demir H, Karakaya C, Ozbek H. Gastroprotective activity of Nigella sativa L oil and its constituent, thymoquinone against acute alcohol-induced gastric mucosal injury in rats. World J Gastroenterol. 2005 Nov 14;11(42):6662-6. doi: 10.3748/wjg.v11.i42.6662. PMID 16425361
- [Background] Seniuk OF, Gorovoj LF, Beketova GV, Savichuk HO, Rytik PG, Kucherov II, Prilutskay AB, Prilutsky AI. Anti-infective properties of the melanin-glucan complex obtained from medicinal tinder bracket mushroom, Fomes fomentarius (L.: Fr.) Fr. (Aphyllophoromycetideae). Int J Med Mushrooms. 2011;13(1):7-18. doi: 10.1615/intjmedmushr.v13.i1.20. PMID 22135899
- [Background] Peterson WL. The role of antisecretory drugs in the treatment of Helicobacter pylori infection. Aliment Pharmacol Ther. 1997 Apr;11 Suppl 1:21-5. doi: 10.1046/j.1365-2036.11.s1.4.x. PMID 9146787
- [Background] Salem EM, Yar T, Bamosa AO, Al-Quorain A, Yasawy MI, Alsulaiman RM, Randhawa MA. Comparative study of Nigella Sativa and triple therapy in eradication of Helicobacter Pylori in patients with non-ulcer dyspepsia. Saudi J Gastroenterol. 2010 Jul-Sep;16(3):207-14. doi: 10.4103/1319-3767.65201. PMID 20616418
- [Background] Poelmans J, Feenstra L, Demedts I, Rutgeerts P, Tack J. The yield of upper gastrointestinal endoscopy in patients with suspected reflux-related chronic ear, nose, and throat symptoms. Am J Gastroenterol. 2004 Aug;99(8):1419-26. doi: 10.1111/j.1572-0241.2004.30066.x. PMID 15307853
- [Background] Poelmans J, Tack J, Feenstra L. Chronic middle ear disease and gastroesophageal reflux disease: a causal relation? Otol Neurotol. 2001 Jul;22(4):447-50. doi: 10.1097/00129492-200107000-00005. PMID 11449097
- [Background] Poelmans J, Feenstra L, Tack J. Determinants of long-term outcome of patients with reflux-related ear, nose, and throat symptoms. Dig Dis Sci. 2006 Feb;51(2):282-8. doi: 10.1007/s10620-006-3126-y. PMID 16534670
- [Background] Schmausser B, Andrulis M, Endrich S, Muller-Hermelink HK, Eck M. Toll-like receptors TLR4, TLR5 and TLR9 on gastric carcinoma cells: an implication for interaction with Helicobacter pylori. Int J Med Microbiol. 2005 Jun;295(3):179-85. doi: 10.1016/j.ijmm.2005.02.009. PMID 16044857
- [Background] Schmausser B, Andrulis M, Endrich S, Lee SK, Josenhans C, Muller-Hermelink HK, Eck M. Expression and subcellular distribution of toll-like receptors TLR4, TLR5 and TLR9 on the gastric epithelium in Helicobacter pylori infection. Clin Exp Immunol. 2004 Jun;136(3):521-6. doi: 10.1111/j.1365-2249.2004.02464.x. PMID 15147355
- [Background] El-Obeid A, Hassib A, Ponten F, Westermark B. Effect of herbal melanin on IL-8: a possible role of Toll-like receptor 4 (TLR4). Biochem Biophys Res Commun. 2006 Jun 16;344(4):1200-6. doi: 10.1016/j.bbrc.2006.04.035. Epub 2006 May 2. PMID 16650380
- [Background] Rakoff-Nahoum S, Paglino J, Eslami-Varzaneh F, Edberg S, Medzhitov R. Recognition of commensal microflora by toll-like receptors is required for intestinal homeostasis. Cell. 2004 Jul 23;118(2):229-41. doi: 10.1016/j.cell.2004.07.002. PMID 15260992
- [Background] Fukata M, Chen A, Klepper A, Krishnareddy S, Vamadevan AS, Thomas LS, Xu R, Inoue H, Arditi M, Dannenberg AJ, Abreu MT. Cox-2 is regulated by Toll-like receptor-4 (TLR4) signaling: Role in proliferation and apoptosis in the intestine. Gastroenterology. 2006 Sep;131(3):862-77. doi: 10.1053/j.gastro.2006.06.017. PMID 16952555
- [Background] Zheng L, Riehl TE, Stenson WF. Regulation of colonic epithelial repair in mice by Toll-like receptors and hyaluronic acid. Gastroenterology. 2009 Dec;137(6):2041-51. doi: 10.1053/j.gastro.2009.08.055. Epub 2009 Sep 2. PMID 19732774
- [Background] Hoogerwerf et al. 2006. Hoogerwerf, W.J., Pasricha, P.J., 2006. Pharmacotherapy of gastric acidity,peptic ulcer and gastroesophageal reflux disease: Goodman and Gilman's.The pharmacological basis of therapeutics. McGraw-Hill, United States, pp.869-882).
- [Background] Wada A, Ogushi K, Kimura T, Hojo H, Mori N, Suzuki S, Kumatori A, Se M, Nakahara Y, Nakamura M, Moss J, Hirayama T. Helicobacter pylori-mediated transcriptional regulation of the human beta-defensin 2 gene requires NF-kappaB. Cell Microbiol. 2001 Feb;3(2):115-23. doi: 10.1046/j.1462-5822.2001.00096.x. PMID 11207625
- [Background] Biragyn A, Ruffini PA, Leifer CA, Klyushnenkova E, Shakhov A, Chertov O, Shirakawa AK, Farber JM, Segal DM, Oppenheim JJ, Kwak LW. Toll-like receptor 4-dependent activation of dendritic cells by beta-defensin 2. Science. 2002 Nov 1;298(5595):1025-9. doi: 10.1126/science.1075565. PMID 12411706
- [Background] Ohara T, Morishita T, Suzuki H, Masaoka T, Nagata H, Hibi T. Pathophysiological role of human beta-defensins 2 in gastric mucosa. Int J Mol Med. 2004 Dec;14(6):1023-7. PMID 15547668